CLINICAL TRIAL: NCT04988555
Title: A Phase 1/2, Open-Label, Dose-Escalation, Dose-Expansion Study of DSP-5336 in Adult Patients With Acute Leukemia and Other Selected Hematologic Malignancies, With and Without Mixed Lineage Leukemia (MLL) Rearrangement or Nucleophosmin 1 (NPM1) Mutation
Brief Title: A Study of DSP-5336 in Relapsed/Refractory AML/ ALL With or Without MLL Rearrangement or NPM1 Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSP-5336-101
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Acute
Keywords: Relapsed or refractory AML; MLLr; Menin; NPM1m; KMT2A
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence | interventions — Azoles; venetoclax; gilteritinib; Azacitidine

STUDY DESIGN:
Intervention Model Description: Bayesian Regression Model for Phase 1 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Phase 1 - Arm A (Experimental): Patients not taking antifungals within 7 days of study entry
  Interventions: Drug: Enzomenib
- Phase 1 - Arm B (Experimental): Patients receiving antifungals that are moderate to strong cytochrome CYP3A4/5 inhibitors (i.e. posaconazole, voriconazole, or fluconazole).
  Interventions: Drug: Enzomenib; Drug: azoles
- Phase 1 - Arm C (Experimental): Patients with MDS
  Interventions: Drug: Enzomenib
- Phase 1 - Arm E (Experimental): Patients with AML
  Interventions: Drug: Enzomenib; Drug: Venetoclax; Drug: Azacitidine (AZA)
- Phase 1 - Arm F (Experimental): Patients with AML
  Interventions: Drug: Enzomenib; Drug: Gilteritinib
- Phase 2 - Arm G (Experimental): R/R AML with MLLr
  Interventions: Drug: Enzomenib
- Phase 2 - Arm H (Experimental): R/R AML with NPM1m
  Interventions: Drug: Enzomenib
- Phase 2 - Arm I (Experimental): R/R ALL with MLLr
  Interventions: Drug: Enzomenib

INTERVENTIONS:
Drug: Enzomenib — DSP-5336 orally
Drug: azoles — Posaconazole, Voriconazole, or Fluconazole
  Arms: Phase 1 - Arm B
Drug: Venetoclax — Venetoclax orally
  Arms: Phase 1 - Arm E
Drug: Gilteritinib — Gilteritinib orally
  Arms: Phase 1 - Arm F
Drug: Azacitidine (AZA) — Azacitidine orally
  Arms: Phase 1 - Arm E

SUMMARY:
A phase 1/2 dose escalation / dose expansion study of Enzomenib (DSP-5336) in adult patients with acute leukemia.

DETAILED DESCRIPTION:
Phase 1 (dose escalation) will determine the recommended Phase 2 dose (RP2D) (i.e. the lowest dose of Enzomenib (DSP-5336), that provides the maximum biologic and clinical effect, or the MTD, whichever is lower) in adult patients with relapsed or refractory AML, ALL, or acute leukemia of ambiguous lineage. Enrollment to the phase 1 portion of the study may be limited to patients with certain genetic abnormalities.

Phase 2 dose-expansion will further evaluate the safety and clinical activity of Enzomenib (DSP-5336) monotherapy in patients with relapsed/refractory AML who have MLLr or NPM1m, and relapsed/refractory ALL who have MLLr.

ELIGIBILITY:
Inclusion Criteria:

Patients in the Phase 1 dose-escalation portion must have a diagnosis of relapsed or refractory AML, ALL or acute leukemia of ambiguous lineage according to World Health Organization (WHO) 2022 classification, or, in the US only, a diagnosis of MDS or MM as determined by pathology review at the treating institution, and whose disease has progressed after available standard therapies known to be active for their AML, ALL, or acute leukemia of ambiguous lineage or, in the US, for MM or MDS.

For patients with MDS (US only):

1. Patients with MDS must have IPSS-R risk categorization of "high" or "very high" at initial diagnosis or at study entry and have bone marrow blasts ≥ 5% (which is the definition of high-risk MDS in this study)
2. Patients with MDS must have relapsed or refractory disease and have exhausted available standard therapies including at least 2 cycles of treatment with HMA

For patients with MM (US only):

1. Have a confirmed diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) 2016 classification (Kumar, 2016) and whose disease has progressed after treatment with a minimum of 3 prior anti-myeloma regimens including a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-CD38 monoclonal antibody (mAb); patients must not be candidates for available therapies with established clinical benefit
2. Have measurable disease as defined in the protocol
3. Meet the laboratory parameters set in the protocol

For patients with relapsed/refractory AML in the venetoclax and azacitidine combination cohort (in countries and sites where permitted):

1. Have MLLr or NPM1m.

   For patients with relapsed/refractory AML in the gilteritinib combination cohort (in countries and sites where permitted):
2. Have MLLr or NPM1m AND any of the following FLT3 mutations: FLT3-ITD, FLT3-TKD/D835 or FLT3-TKD/I836.

Patients in the Phase 2 dose expansion portion of the study must have a confirmed diagnosis of relapsed AML or ALL as determined by pathology review at the treating institution, and who have ≥5% blasts by morphologic assessment in the bone marrow and failed available standard therapies known to be active for their AML (Arm G and H) or ALL (Arm I). If the primary disease is a transformation from MDS or other hematologic malignancies, patients need to receive available standard therapies for acute leukemia before enrolling this trial. Participants who are candidates for stem cell transplantation must have been offered this therapeutic option. Patients with extramedullary disease or peripheral blasts as the only manifestation of relapse are not eligible.

1. Patients must not have had prior exposure to a menin inhibitor
2. Patients for Arms G and H are limited to a total of 3 prior lines of therapy, with induction chemotherapy, consolidation chemotherapy, and stem cell transplantation with or without subsequent maintenance treatment considered to be 1 line.
3. Have a documented KMT2A (MLL)-fusion for Arm G and I or NPM1 mutation for Arm H assessed at relapse or immediately prior to the determination of refractory status. For Arms G and I, KMT2A genetic alterations other than fusions (eg, KMT2A-PTD, amplification, point mutation) are not permitted.
4. Be > 18 years of age. For countries and sites where approved, for DSP-5336 monotherapy, acute leukemia patients ≥12 years of age who weigh ≥40 kg may be enrolled.
5. ECOG < 2; For Phase 2 only, patients must have an ECOG performance status 0 or 1.
6. For monotherapy, WBC below 30,000/μ. For the combination arms, WBC count must be below 25,000/uL at enrollment and prior to starting treatment. (Hydroxyurea and steroids for cytoreduction purposes are allowed prior to enrollment and during study treatment)
7. Clearance of creatinine (CLcr) level ≥ 50 ml/min, assessed by the Cockcroft-Gault formula
8. Total bilirubin ≤1.5 the upper limit of normal (ULN) (or ≤2.0 ULN for patients with known Gilbert's syndrome)
9. Aspartate aminotransferase (AST) ≤3.0 times ULN
10. Alanine aminotransferase (ALT) ≤3.0 times ULN
11. Any prior treatment-related toxicities resolved to ≤Grade 1 prior to enrollment, with the exception of ≤Grade 2 alopecia or neuropathy.
12. Be willing to attend study visits as required by the protocol
13. Have an estimated life expectancy ≥3 months, based on the investigator's assessment
14. Females of childbearing potential must have a negative serum pregnancy test.
15. Must agree to use a highly effective contraception method or 2 acceptable methods of birth control (each partner must use one method) or use prevention of pregnancy measures (ie, agreement to refrain completely from heterosexual intercourse) during the study and for 6 months (for females and males alike) after the last dose of study drug, if male or female patient is of child-producing potential

    For sites in Japan only: Implantable hormonal contraceptives, a diaphragm with spermicide, cervical cap with spermicide and contraceptive sponge (spermicide is already in the contraceptive sponge) included in the barrier contraceptive method are not approved and cannot be used in Japan.
16. Have AML/ALL/MDS/MM bone marrow material suitable for genomic analysis of AML,ALL, MDS, or MM genetic alterations. Note: If a bone marrow material is insufficient, an alternative suitable tissue (ex: peripheral blood) must be provided.

Exclusion Criteria:

1. Has a left ventricular ejection fraction (LVEF) <50%, as determined by ECHO
2. Histological diagnosis of acute promyelocytic leukemia
3. Received systemic calcineurin inhibitors within 2 weeks prior to the first dose of DSP 5336
4. Have abnormal ECGs at screening that are clinically significant, such as (QTc >480 msec, with QTc corrected according to Fridericia's formula (QTcF). Note: In case of bundle branch block, QT interval correction can be performed.
5. Has an active anduncontrolled, bacterial, viral, or fungal infection requiring parenteral therapy. Note: Patients must be afebrile with negative blood cultures at least 72 hours prior to Cycle 1 Day 1.
6. Receives concurrent sensitive substrates with a narrow safety window or strong inhibitors or inducers of CYP3A4/5, including specifically: ketoconazole, isavuconazole and itraconazole. Other antifungals that are used as standard of care to prevent or treat infections are permitted. If a patient is on one of the excluded azole class antifungals, he/she can be taken off or switched to a permitted azole 7 or more days prior to first dose, then the patient could be allowed on study (Arm B) with approval of the medical monitor.
7. Received immunotherapy, including tumor vaccines and checkpoint inhibitors, within 42 days prior to the first dose of DSP-5336
8. Had major surgery within 28 days prior to the first dose of DSP-5336
9. Has active central nervous system leukemia. Patients with a history of any CNS leukemia involvement are excluded from Phase 2 Arms G and H.
10. Underwent HSCT or chimeric antigen receptor cell (CAR-T) therapy or other modified T-cell therapy within 60 days prior to the first dose of DSP-5336. Patients who have received >1 prior HSCT are excluded from Phase 2 Arms G and H.
11. Received a donor lymphocyte infusion within 28 days prior to the first dose of DSP-5336, or receiving immunosuppressive therapy post-HSCT at the time of screening, or with clinically active GVHD or GVHD requiring active medical intervention other than the use of topical steroids for ongoing cutaneous GVHD
12. Received antineoplastic agents (except hormonal therapies as adjuvant maintenance for breast or prostate cancers if a patient is taking before starting study treatment, and hydroxyurea given for controlling blast cells) or other investigational treatment within 14 days or 5 half-lives, whichever is shortest, prior to the first dose of DSP-5336
13. In the opinion of the treating investigator, have any concurrent conditions that could pose an undue medical hazard or interfere with interpretation of study results
14. Have a known detectable viral load for human immunodeficiency virus or hepatitis C, or evidence of hepatitis B surface antigen, all being indicative of active infection.

    For sites in Japan, Taiwan, and Korea only: Hepatitis B core (HBc) antibody or hepatitis B surface (HBs) antibody test should be performed if HBsAg is negative. If HBc antibody or HBs antibody test is positive, HBV DNA quantification test should be performed to confirm that HBV DNA is negative.
15. Have severe dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally, including the inability to swallow oral medication
16. Have cognitive, psychologic, or psychosocial impediment that would impair the ability of the patient o receive therapy according to the protocol, or adversely affect the ability of the patient to comply with the informed consent process, protocol, or protocol-required visits and procedures
17. Are pregnant or breastfeeding or planning to become pregnant. Note: Patients who are breastfeeding may be enrolled if they interrupt breastfeeding prior to the first dose of any study drugs and do not feed the baby with breast milk expressed after receiving the first dose of any study drugs. Breastfeeding should not be resumed for at least 6 months after the last dose of study drug
18. Have any history or complication of interstitial lung disease (for sites in Japan in Phase 1 dose escalation only).

    For clinical sites in the EU, have a history of Grade ≥ 2 drug-induced interstitial lung disease or Grade ≥ 2 non-infectious pneumonitis within 6 months of starting study treatment.
19. Have a history of Torsades de Pointes
20. Received systemic calcineurin inhibitors within 4 weeks prior to the first dose of DSP-5336
21. Have plasma cell leukemia (>2.0 x 109 /L plasma cells in blood by standard differential) (for patients with MM only)
22. For patients intending to enroll into the combination cohort with gilteritinib: Patients must be gilteritinib-naïve or sensitive and have not received a FLT3 inhibitor in the relapsed refractory setting (prior FLT3 inhibitor in front line therapy is allowed)
23. Have a known intolerance of hypersensitivity reaction to components of the investigational medicinal product
24. Patients with LDH >500 U/L (>8.3 µkat/L) are excluded from Phase 2 Arms G and H

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase I Assess the safety and tolerability of DSP-5336 in relapsed/refractory AML, ALL or acute leukemia of ambiguous lineage | Approximately 2 months after first dose
  Occurrence of DLTs and frequency, duration and severity of TEAEs and SAEs assessed by NCI CTCAE v 5.0
Phase I Determine the RP2D based on lowest dose of DSP-5336 that provides the maximum biologic and clinical effect, or the MTD, whichever is lower. | Approximately 2 months after first dose
  Occurrence of DLTs and frequency, duration and severity of TEAEs and SAEs, plasma concentration-time profiles, changes in expression levels of biomarkers (gene expression levels).
Phase 2 To evaluate clinical activity of DSP-5336 in adult patients with Relapsed /refractory AML who have MLL (KRMa gene rearrangement or NPM1 gene mutation) | Approximately 6 months after first dose
  Occurrence of CR(MRD-); CR; CRh; CRi; PR; MLFS; CR(MRD-) + CR; CR(MRD-) + CR + CRh; OR (=CR(MRD-) or CR or CRi or MLFS or PR); DOR; time to response; time to CR; TI; OS; EFS; RFS

SECONDARY OUTCOMES:
Phase I Preliminary clinical activity of DSP-5336 in adult patients with AML or ALL | Approximately 6 months after first dose
  Disease response as assessed by ELN 2017 criteria
2. Phase 2 To further assess safety and tolerability of DSP-5336 in adult patients with Relapsed /refractory AML | Approximately 2 months after first dose
  Frequency, duration, and severity of TEAEs and SAEs assessed by NCI CTCAE v 5.0

CONTACTS AND LOCATIONS:
Locations (92):
- United States (29):
  - Hoag Family Cancer Center, Newport Beach, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami, Miami, Florida
  - Northwestern, Chicago, Illinois
  - Sibley Memorial Hospital, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Main Center, Baltimore, Maryland
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Atlantic Health, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - UNC Hospital, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Atrium Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Sidney Kimmel Comprehensive Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - MDACC, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Belgium (4):
  - ZNA Cadix, Antwerp
  - UZ Ghent, Ghent
  - University Hospitals Leuven, Leuven
  - AZ Delta, Roeselare
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta, Edmonton
- France (11):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nice - Hôpital l'Archet 1, Nice
  - Hopital Saint-Louis, Paris
  - CHU Bordeaux, Talence
  - Institut Gustave Roussy, Villejuif
- Italy (7):
  - Alma Mater Studiorum University Of Bologna, Bologna
  - Ospedale Policlinico San Martino, IRCCS, Genoa
  - IRCCS istituto Romagnolo per lo studio dei tumori "Dino Amadori", Meldola
  - Istituto Oncologico Veneto (IOV), IRCCS, Padua
  - Università degli Studi di Perugia, Perugia
  - PU A. Gemelli, Università Cattolica del Sacro Cuore, Rome
  - Universita' Degli Studi Di Torino, Turin
- Japan (11):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Osaka University Hospital, Osaka
- National University Cancer Institute, Singapore, Singapore
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul
- Spain (11):
  - Hospital General Universitario De Albacete, Albacete
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Fundacion Instituto de Investigacion Marques de Valdecilla, Cantabria
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitario De Gran Canaria Dr. Negrin, Las Palmas
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (9):
  - University Hospitals of Birmingham Centre for Clinical Hematology, Birmingham
  - Bristol Hematology & Oncology Centre, Bristol
  - King's College Hospital, London
  - Sarah Cannon Research Institute, London
  - University College London Hospitals NHS Foundation Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Churchill Hospital Oxford, Oxford
  - University Hospitals of North Midlands NHS Foundation Trust, Stoke-on-Trent
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Undecided